CLINICAL TRIAL: NCT00244504
Title: The Effects of Small Doses of Moxonidine in Patients Undergoing Vascular Surgery
Brief Title: Moxonidine in Patients Undergoing Vascular Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped after pre-definied interim analysis because of no effects
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: PD Dr. M. Filipovic, Co-Head of Cardiothoracic Anaesthesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 158/01
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Cardiac Disease; Vascular Surgery
MeSH Terms: conditions — Heart Diseases | interventions — moxonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): moxonidine group
  Interventions: Drug: moxonidine
- II (Placebo Comparator): placebo group
  Interventions: Drug: moxonidine

INTERVENTIONS:
Drug: moxonidine — moxonidine 0.2 mg/d starting the morning of surgery until day 4 after surgery
  Other Names: Physiotens

SUMMARY:
Investigating the perioperative effect of moxonidine. In a randomized double-blind fashion, patients undergoing vascular surgery will receive moxonidine 0.2 mg or placebo from the day before surgery until day 4 after surgery. Holter-EKG for 48 h, starting just before surgery. Repeated 12-lead EKG, measurements of Troponin I and BNP, clinical visitations, follow-up interviews at 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* abdominal aortic or peripheral vascular surgery

Exclusion Criteria:

* unstable angina,
* severe symptomatic heart failure (NYHA IV)
* systolic blood pressure at rest < 100 mmHg
* bradycardia (<50/min)
* higher grade AV heart block
* creatinine clearance < 30 ml/min
* pregnancy
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2002-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
over-all mortality | 30 days and 12 months

SECONDARY OUTCOMES:
Ischemia detected by Holter-ECG ST alterations or troponin T elevation | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Filipovic, PD Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University hospital, Basel, CH, Switzerland

REFERENCES:
- [Derived] Bolliger D, Seeberger MD, Lurati Buse GA, Christen P, Gurke L, Filipovic M. Randomized clinical trial of moxonidine in patients undergoing major vascular surgery. Br J Surg. 2007 Dec;94(12):1477-84. doi: 10.1002/bjs.6012. PMID 17968979